CLINICAL TRIAL: NCT02539355
Title: Diet and Metabolic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Mario Kratz, Associate Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCI2P30CA015704; CCSG Y39 Pilot: Kratz, M (Other Grant/Funding Number: CCSG)
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Resistance; Diabetes; Cancer; Obesity; Inflammation
Keywords: Insulin resistance; Diabetes; Cancer; Obesity; Inflammation
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Neoplasms; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet A (Active Comparator): Standard Healthy Diet (Diet A)
  Interventions: Other: Diet A
- Diet B (Experimental): Alternative Test Diet (Diet B)
  Interventions: Other: Diet B

INTERVENTIONS:
Other: Diet A — 12-week diet
  Arms: Diet A
Other: Diet B — 12-week Diet
  Arms: Diet B

SUMMARY:
Obesity is a risk factor for several common cancers, including those of the breast, colon, liver, and pancreas. Proposed molecular links between obesity and these types of cancer include systemic inflammation, hyperinsulinemia, and changes in the serum concentrations of sex steroid hormones and adipokines. All of these are strongly linked to low-grade chronic inflammatory processes in expanded adipose tissue. The objective of this proposal is to test the hypothesis that adipose tissue inflammation can be reduced by the foods we eat.

DETAILED DESCRIPTION:
Overweight or obese individuals with evidence of insulin resistance will be enrolled, until 16 have completed all study procedures. Enrolled subjects will be randomized to follow one of two healthy diets for 12 weeks to determine how each diet affects inflammation in the body and sugar and insulin levels in the blood.

We will address the following specific aims:

Primary specific aim: To investigate whether the consumption of either diet reduces the metabolic activation of adipose tissue macrophages (ATM) as assessed by quantifying the ATM cell surface expression (relative mean fluorescence intensity, rMFI) of the metabolic activation markers, CD36 and ABCA1.

Secondary specific aim 1: To compare how each of the study diets affects endpoints downstream of metabolic activation of ATM, specifically (a) adipose tissue expression of the key pro-inflammatory cytokines tumor necrosis factor α (TNFα) and interleukins (IL)-1 beta and 6; (b) adipose tissue expression of the key anti-inflammatory adipokine, adiponectin; (c) systemic insulin sensitivity, as assessed by the Matsuda-DeFronzo Insulin Sensitivity Index (ISI), based on a 3-hour frequently sampled oral glucose tolerance test (FS-OGTT); and oral glucose tolerance, as assessed by measuring the total area-under-the-curve glucose in the FS-OGTT.

Secondary specific aim 2: To compare the impact of each of the study diets on low-grade chronic systemic inflammation, as assessed by measuring the concentrations of high sensitivity C-reactive protein (hsCRP), IL-6, and total adiponectin in fasting plasma.

Secondary specific aim 3: To assess dietary adherence in the two dietary intervention groups. Dietary adherence will be measured by a dietary adherence score (separately for each diet), based on repeated 4-day diet records completed by all participants in the study.

Because all of our study endpoints are thought to be linked to the gut microbiota, and because the effects of diet may be mediated through changes in the gut microbiota, we will also collect stool samples from all participants before and after completing the study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 28 kg/m2
* Homeostasis model assessment insulin resistance (HOMA-IR) index > 2.0
* Body weight within 10% of weight 3 months before starting the study
* Able to come to the FHCRC Prevention Center for one 1-hour pre-study visit and two clinic visits of ~4.5 hours duration each
* Able and willing to attend bi-weekly dietary group counseling sessions at FHCRC during the 12-week intervention period
* Willingness and ability to follow the dietary regimen
* Able to complete repeated 3-day food records before and during the dietary intervention.
* Willingness to maintain usual lifestyle habits (other than diet) throughout the study (e.g., physical activity habits)
* Ability to understand, speak, and write in English
* Ability to provide informed written consent

Exclusion Criteria:

* Any previous or current use of antidiabetic medications or insulin
* Presence or history of major chronic inflammatory or autoimmune disease (e.g., lupus, rheumatoid arthritis, Hashimoto's thyroiditis, inflammatory bowel disease, celiac disease, multiple sclerosis), malabsorption syndromes, or diseases of the liver, thyroid, or kidneys (stage IV or later chronic kidney disease)
* Food allergies or intolerances against major study foods
* Intake of drugs likely to interfere with study endpoints, including corticosteroids and anabolic steroids, hormone replacement therapy, NSAIDS (more than 3 times per week and/ or more than 600 mg per day), warfarin (within 3 months of starting the study), antibiotics or probiotics (within 2 weeks of starting the study)
* Presence or recent history of anemia (within 3 months of starting the study)
* Participation in another study that includes an intervention of any kind or a blood draw >300 mL over 3 months
* Alcohol intake > 2 drinks per day
* Use of tobacco products, eCigarettes, or recreational drugs on more than 2 days per month
* Current or recent (within 12 months of starting the study) pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in adipose tissue macrophage cell surface expression of metabolic activation marker CD36 as measured by relative mean fluorescence intensity | Change between beginning (day 1) and end (week 12) of the study diet period.
  As measured by relative mean fluorescence intensity (rMFI) on abdominal subcutaneous adipose tissue macrophages
Change in adipose tissue macrophage cell surface expression of metabolic activation marker ABCA1 as measured by relative mean fluorescence intensity (rMFI) | Change between beginning (day 1) and end (week 12) of the study diet period.
  As measured by relative mean fluorescence intensity (rMFI) on abdominal subcutaneous adipose tissue macrophages

SECONDARY OUTCOMES:
Change in adipose tissue expression of the key pro-inflammatory cytokine, tumor necrosis factor α (TNFα) assessed by qPCR | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by qPCR on whole abdominal subcutaneous adipose tissue
Change in adipose tissue expression of the key pro-inflammatory cytokine, interleukin-6 (IL-6) assessed by qPCR | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by qPCR on whole abdominal subcutaneous adipose tissue
Change in adipose tissue expression of the key pro-inflammatory cytokine, interleukin-1 beta (IL-1beta) assessed by qPCR | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by qPCR on whole abdominal subcutaneous adipose tissue
Change in adipose tissue expression of the key anti-inflammatory adipokine, adiponectin assessed by qPCR | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by qPCR on whole abdominal subcutaneous adipose tissue
Change in systemic insulin sensitivity assessed by the Matsuda-DeFronzo Insulin Sensitivity Index | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by the Matsuda-DeFronzo Insulin Sensitivity Index (ISI) based on a 3-hour frequently sampled oral glucose tolerance test (FS-OGTT)
Change in oral glucose tolerance assessed by measuring total area under the curve glucose in the FS-OGTT | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by measuring total area under the curve glucose in the FS-OGTT
Change in fasting plasma C-reactive protein assessed by immunonephelometry | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by immunonephelometry
Change in fasting plasma IL-6 assessed by high-sensitivity ELISA | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by high-sensitivity ELISA
Change in fasting plasma total adiponectin assessed by ELISA | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by ELISA

OTHER OUTCOMES:
Dietary adherence to prescribed 12-week diet assessed by dietary compliance score | Assessed at the end of the study (week 12).
  Assessed by dietary compliance score, based on data from repeated 4-day dietary records
Changes in gut microbiota assessed by stool sample analysis | Change between beginning (day 1) and end (week 12) of the study diet period.
  Assessed by stool sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States